CLINICAL TRIAL: NCT00287274
Title: Impact of Computerized Physician Order Entry on Medication Prescription Errors in the Intensive Care Unit: a Controlled Cross-Sectional Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2004/002
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Medication Errors; Patient Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: computerized physician order entry

SUMMARY:
Device: computerized physician order entry.

We wanted to investigate if the introduction of a computerized intensive care unit system reduced the incidence and severity of medication prescription errors (MPEs). A prospective trial was conducted during 5 weeks in a paper-based unit versus a computerized unit. The registration of different classes of MPEs was done by a clinical pharmacist. An independent panel evaluated the severity of MPEs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the Surgical Intensive Care Unit

Exclusion Criteria:

* Adult Patients admitted to other units
* Pediatric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2004-03; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
To compare the the incidence and severity of medication prescription errors between a CPOE unit and a paper-based unit at completion of the study.

SECONDARY OUTCOMES:
Description of MPEs in both units at completion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Colpaert, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Result] Colpaert K, Claus B, Somers A, Vandewoude K, Robays H, Decruyenaere J. Impact of computerized physician order entry on medication prescription errors in the intensive care unit: a controlled cross-sectional trial. Crit Care. 2006 Feb;10(1):R21. doi: 10.1186/cc3983. PMID 16469126
- See also: Website University Hospital Ghent — http://www.uzgent.be